CLINICAL TRIAL: NCT03370978
Title: The Role of Text Messaging in Follow-up Appointments for Patients Discharged From the Emergency Department
Brief Title: Text Messaging Follow-up From ED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started as no longer novel
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Brooks Obr, Principal Investigator, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201607734
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Text Messaging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Messaging (Experimental): Receives text messages to remind of upcoming follow-up appointment with primary care doctor. Also provides opportunity for subjects to text ED staff for follow-up care concerns or to reschedule primary care appointment.
  Interventions: Behavioral: Text Messaging
- Usual Care (No Intervention): Received usual care including follow-up phone calls if clinically indicated.

INTERVENTIONS:
Behavioral: Text Messaging — To communicate with intervention patients after discharge from the ED, we will use a bidirectional text messaging service provided by another physician's research group within the University of Iowa. The nurse navigator will enter the patient's study identification number, first and last name and cell phone onto a secure study website established by this research group.
  Patients will, as previously mentioned, have had their cell phone number tested in the text messaging system prior to leaving the Emergency Department (this includes the control group).
  Patient's will receive a text message 3 days, and 1 day, prior to their scheduled follow-up appointment with Family Medicine (this appointment having been scheduled through the Emergency Department Nurse Navigators). Each text message will remind the patient of the date/time of their appointment, and provide them a link containing a map with the location of their appointment.
  Arms: Text Messaging

SUMMARY:
Ensuring follow-up for patients after discharge from the emergency department (ED) has long been a concern for ED care providers. The current technology of text messaging may be able to assist us in improving follow-up rates. In addition, having a quick and easy communication tool to be in touch with providers may improve overall patient satisfaction. This study is designed to evaluate the usage of text messaging to improve follow-up appointment compliance from the Emergency Department. In this study, a prospective randomized controlled trial (RCT) will be performed (involving patients scheduled by Emergency Department Nurse Navigators to follow up with Family Medicine) in which patients will be randomized to a texting appointment reminder versus standard-of-care (no texting reminder) group. Texted patients will receive reminders 3 days and 1 day prior to their follow-up appointment. In addition, the patients will have the ability to text back-and-forth with the Nurse Navigators in order to ask questions/request clarification if needed. Chart review will be performed of both groups to evaluate the number of follow-up appointments that patients attended versus rescheduled versus did not attend/reschedule. These values will then be compared to the retrospective chart review previously performed to evaluate for non-inferiority of text messaging as a means of improving patient attendance at follow-up appointments.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Able to read, write and communicate in English - English as the primary language
3. Has a phone with capabilities for text messaging
4. Identifies oneself as someone who is comfortable with text messaging.
5. To follow-up with Family Medicine as outpatient (Scheduled through Emergency Department Nurse Navigators).
6. Evaluated in the University of Iowa Hospitals and Clinics Emergency Department

Exclusion Criteria:

1. Absence of one or more inclusion criteria
2. Not able to provide informed consent or participate due to limited decision-making ability.
3. Prisoner
4. Previously has followed with the University of Iowa Hospitals and Clinics Family Medicine (i.e., would not be a "new" patient establishing care).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Attending Primary Care Appointment | Less than 6 months
  Attending appointment versus rescheduling versus not showing

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared